CLINICAL TRIAL: NCT03476200
Title: Hair Cortisol Concentrations as Indicator of Efficacy of Cognitive Behavioral Therapy
Brief Title: Efficacy of Cognitive Behavioral Therapy and Hair Cortisol Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María Ángeles García León, Principal Investigator, Universidad de Granada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STR2017
Record Dates: First submitted 2018-03-11; First posted 2018-03-23 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Cognitive Therapy; Control
Keywords: Cognitive Behavioral Therapy; Hair Cortisol; Hypothalamic Pituitary Adrenal Axis; Stress; Psychopathology
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy consisting of fourteen weekly group sessions, one hour and a half each, directed by two clinical psychologist.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Control Group (No Intervention): Control Group with no intervention.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The intervention consist of 14 weekly group meetings lasting 1.5 or 2 h. Groups are made up of 10 patients. Each group session follow a structured format and consisted of the following elements: introduction to the session, discussion of homework, group discussion and the development of new coping skills. The sessions deal with the following: concept of stress, cognitive restructuring, alternative thought control strategies, relaxation techniques, training in social skills, training in social skills and humour and optimism as coping strategies.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Stress is considered as a risk factor for physical and mental health. For this reason, interventional programs focused on stress management have been developed. These programs have proven to be efficacious modifying emotional variables and psychopathological symptoms. However, there are no studies showing how these interventions modify objective measures of stress. For example, measures reflecting Hipotalamic-Pituitary-Adrenal (HPA) axis activity, the main system involved in the stress response. The activity of HPA axis is also altered by illness and psychopathology. Hair cortisol technique allows for changes assessment of HPA axis activity during months. Therefore, hair cortisol may be considered as an useful tool to measure changes of emotional variables related to stress in the long term. This measure of change over time of HPA axis activation together with related emotional variables assessment could be useful to evaluate the efficacy of interventional programs. For this reason, the aim of this research is to assess the effects of a cognitive-behavioral treatment (CBT) on perceived stress, resilience, worries, psychopathology and HPA axis activity through hair cortisol analysis.

ELIGIBILITY:
Inclusion Criteria:

* Member of University of Granada, complete dominance of spanish, high levels of perceived stress.

Exclusion Criteria:

* Psychopathology, being under psychological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in "Connor and Davidson Resilience Scale" (CD-RISC) scores. | Three measures: at the beginning of the study, at three months (when the stress program is finished) and at three months follow up (since the end of the stress program).
  The scale measures resilience as the ability to successfully cope with stress, punctuations range from 0 to 100, higher scores indicate higher levels of resilience.
Changes of Hair Cortisol Levels | Three measures: at the beginning of the study, at three months (when the stress program is finished) and at three months follow up (since the end of the stress program).
  The technique measures hypothalamic-pituitary-adrenal axis activation during the last three months, higher levels indicate higher activation of HPA axis.

SECONDARY OUTCOMES:
Changes in "The Cohen Perceived Stress Questionnaire" (PSQ) scores. | Three measures: at the beginning of the study, at three months (when the stress program is finished) and at three months follow up (since the end of the stress program).
  The questionnaire measures perceived stress during the last month, the punctuations range from 0 to 56, higher scores indicate higher levels of perceived stress.
Changes in "The Stress Vulnerability Inventory" (SVI) scores. | Three measures: at the beginning of the study, at three months (when the stress program is finished) and at three months follow up (since the end of the stress program).
  This Inventory measures the predisposition to be affected by perceived stress, the punctuations range from 0 to 22, higher scores indicate more vulnerability to stress.
Changes in "Symptoms Checklist-90-Revised" (SCL-90-R) scores. | Three measures: at the beginning of the study, at three months (when the stress program is finished) and at three months follow up (since the end of the stress program).
  This scale is a screening tool to measure psychopathological symptoms, it is formed by 9 sub scales (each sub scale refers to one type of psychopathology), all the sub scales scores range from 5 to 99, considering 70 as a clinical punctuation.
Changes in "Penn State Worry Questionnaire" (PSWQ) scores. | Three measures: at the beginning of the study, at three months (when the stress program is finished) and at three months follow up (since the end of the stress program).
  The questionnaire measures the level of permanent worries and the cognitive components of anxiety, the scores range from 16 to 80, higher punctuations indicate higher levels of worries.
Changes in "Life Orientation Test Revised" (LOT-R) scores. | Three measures: at the beginning of the study, at three months (when the stress program is finished) and at three months follow up (since the end of the stress program).
  This test measures dispositional optimism, scores range from 0 to 40, higher punctuations indicate higher levels of optimism.
Changes in "Nottingham Health Profile" (NHP) scores. | Three measures: at the beginning of the study, at three months (when the stress program is finished) and at three months follow up (since the end of the stress program).
  This scale measures perceived state of health, it has 6 sub scales (each corresponds to one health dimension), all the sub scales scores range from 0 to 1, higher punctuations indicates poorer state of health on that dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Peralta-Ramírez, Prof, Study Director — Universidad de Granada
Locations (1):
- Department of Personality, Assessment and Psychological Treatment, University of Granada, Granada, Spain